CLINICAL TRIAL: NCT05323097
Title: Drowning-related Out-of-hospital Cardiac Arrest in Denmark: A Six-year Registry-based Study
Brief Title: Drowning-related OHCA in Denmark: A Six-year Registry-based Study
Status: Completed | Type: Observational
Sponsor: Prehospital Center, Region Zealand (Other)
Responsible Party: Principal Investigator, Niklas Breindahl, Medical Doctor, PhD-student, Prehospital Center, Region Zealand
Other Study IDs: DROWN_OHCA
Record Dates: First submitted 2022-03-25; First posted 2022-04-12 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Drowning; Out-Of-Hospital Cardiac Arrest
Keywords: Drowning; Out-Of-Hospital Cardiac Arrest; Water; Register study; Retrospective
MeSH Terms: conditions — Drowning; Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Drowning-related OHCA: Drowning-related OHCA: YES
  Interventions: Other: Drowning-related OHCA
- All other OHCA: Drowning-related OHCA: NO

INTERVENTIONS:
Other: Drowning-related OHCA — Drowning-related out-of-hospital cardiac arrest (OHCA): YES
  Groups: Drowning-related OHCA

SUMMARY:
Within a six-year period from 2016-2021, this retrospective cohort study aims to: 1) report the national incidence of drowning related OHCA's among cases attended by the Danish Emergency Medical Services (EMS), 2) assess survival defined as return of spontaneous circulation (ROSC) on scene, by hospital admission and 30-day survival.

Furthermore, aspects associated with better outcome are evaluated including actions taken by EMS-personnel and laypersons, geographical localization, type of activity, witnessed event, EMS response times, bystander CPR, initial rhythm, use of defibrillator, airway devices, pre-hospital medication, and patient demographics.

This can potentially result in recommendations towards certain educative, preventative, rescue, or treatment strategies to reduce OHCA from drowning.

DETAILED DESCRIPTION:
Introduction

Preventing drowning accidents is of great interest, as a large proportion of drowning events can be avoided by proper educative and targeted preventive measures. Yet, effective educative, preventative, rescue and treatment interventions to reduce fatal drowning events require accurate, reliable and sufficient data to be scientifically analysed. However, the complexity of the disease, various drowning terminology, definitions, and an inappropriate classification of drowning events even in high-income countries possess a great challenge when trying to gather sufficient data.

Currently, drowning is a major cause of mortality worldwide, and a leading cause of cardiac arrest in children and adolescents. Even in highly developed countries, the incidence of drowning is highest among children less than 5 years of age and in young adults between 15 and 24 years of age. The duration of submersion plays a key role in determining the outcome from drowning, as submersion exceeding 10 minutes is associated with poor outcome. Furthermore, drowning leading to hypoxic cardiac arrest is a reversible cause that can be treated. Therefore, bystanders, trained rescuers (e.g., trained lifeguards) and EMS personnel play a critical role in the initial attempts at rescue and resuscitation to prioritize oxygenation and ventilation.

Yet, research on out-of-hospital cardiac arrest (OHCA) due to drowning is limited, and under reporting contributes significantly to misunderstanding of the process of drowning. This leads to a potential for improvement, which requires first and foremost clarification of the most obvious causes and risk factors associated with OHCA from drowning following recommended guidelines for uniform reporting of data from drowning.

Thus, within a six-year period, this study aims to: 1) report the national incidence of drowning related OHCA's among cases attended by the Danish Emergency Medical Services (EMS), 2) to assess survival defined as return of spontaneous circulation (ROSC) at any time followed by status at admission and 30-day survival.

Furthermore, aspects associated with better outcome are evaluated including actions taken by EMS-personnel and laypersons, geographical localization, type of activity, witnessed event, EMS response times, bystander CPR, initial rhythm, use of defibrillator, airway devices, pre-hospital medication, and patient demographics.

This can potentially result in recommendations towards certain educative, preventative, rescue, or treatment strategies to reduce OHCA from drowning.

Methods

Terminology: Drowning is defined by the WHO in 2002 as "the process of experiencing respiratory impairment from submersion or immersion in liquid". Submersion is the situation where the victim's entire body, including the airway, goes below the surface of the liquid. Immersion is to be covered in water, and for drowning to occur, usually at least the face and airway are immersed. If the victim is rescued at any time, the process of drowning is interrupted, which is termed a nonfatal drowning. If the person dies at any time because of drowning, this is termed a fatal drowning. Any submersion or immersion event without evidence of respiratory impairment is considered a water rescue and not a drowning. Terms such as "near drowning", "dry or wet drowning", "secondary drowning", "active and passive drowning", and "delayed onset of respiratory distress" should be avoided.

Setting: In 2016 the Danish Emergency Medical Services (EMS) introduced a nationwide electronic medical reporting system recording all following cases of OHCA in which a resuscitative attempt was initiated in the Danish Cardiac Arrest Registry. Together with a manual validation process, this electronic system is the cornerstone in the Danish out-of-hospital cardiac arrest (OHCA) registry, a solid base for identification and verification of OHCA. Because of the changeover a validation team manually processed all records extracted from the electronic medical records. This ensured high-quality data from the approximately 5,400 annually registered OHCA in Denmark, within the period from 2016 to 2018. From the direct registration and later manual verification, several additional data sources were coupled with each registered OHCA (e.g., survival, initiation of bystander CPR and potential drowning accident).

This enables the possibility for advanced text searching in the entire pre-hospital medical record for cases with OHCA. In a pilot-study performed at Zealand EMS in 2019, a feasible and efficient method for identifying OHCA from foreign body airway obstruction was developed, based on identification of trigger-words in the electronic medical record.

Identification of fatal drowning accidents: During the manual validation of OHCA in the changeover period, 211 cases were flagged as drowning accidents. However, the obstacle of manual verification across EMS regions persists and further data cleansing and revised search-strings are needed to provide high-quality data. Therefore, the investigators will identify trigger-words in the 211 electronic reports from the initial screening by manually reading through the medical records. A text-string based on these trigger-words will be structured and fed into a text-search algorithm able to search note-fields within the electronic medical records. When searching the electronic medical records from the OHCA register, the algorithm will return several records, consisting of OHCA presumably caused by drowning. However, the initial search alone will miss some of the manually registered OHCA caused by drowning and conversely, non-fatal drowning accidents not registered in the Danish Cardiac Arrest Registry will also be identified from the search, which need to be excluded in this research project. After a manual review of the specified reports, new trigger-words will be added to the search-string to include reports not identified during the initial manual registration ultimately leading to a revised text-string. This iterative process will be performed until no new reports appear, and the investigators will have identified the final number of OHCA presumably caused by drowning. The remaining four regions have all pledged data permission and agreed to initiate the study when funding has been acquired.

Perspectives: This study provides novel information regarding OHCA related to drowning; the descriptive statistics provides relevant data based on a reviewed, high-quality database. Furthermore, this study will enable targeted campaigns aimed at increasing survival from OHCA caused by drowning, targeting preventative actions in means of educating the public, creating awareness, increasing signage and potentially allocating lifeguards to high-risk areas, or establishing public lifeguard training and bystander initiatives.

ELIGIBILITY:
Inclusion Criteria:

* Out-of-hospital cardiac arrest (OHCA)

Exclusion Criteria:

* Obvious clinical signs of irreversible death (decapitation, decomposition, postmortem lividity, postmortem rigidity)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All Danish citizens with out-of-hospital cardiac arrest in the period from 2016-2021.
Sampling Method: Probability Sample
Enrollment: 31200 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
30-day survival | 30-day after OHCA
  Alive or Dead 30 days after the event.

SECONDARY OUTCOMES:
Annual incidence and survival rates of drowning-related OHCA per 100,000 from 2016-2021 | Annually from 2016-2021 (at the end of the year)
  Stratified by the most obvious causes and risk factors following recommended guidelines for uniform reporting of data from drowning including precipitating event, geographical localization, and type of activity
Map of drowning-related OHCA in Denmark from 2016-2021 | 5-year period from 2016-2021
  Showing a map of geographical localization of drowning-related OHCA in Denmark in the study period indicating 30-day mortality and survival
Survival status at hospital admission | At hospital admission within 24 hours after admission
  ROSC (unconscious) at hospital admission, ROSC (conscious) at hospital admission, Ongoing CPR at hospital admission, Dead at hospital admission

CONTACTS AND LOCATIONS:
Overall Officials: Niklas Breindahl, MD, Principal Investigator — Prehospital Center, Region Zealand, Denmark
Locations (1):
- Prehospital Center, Næstved, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: Yes
The study protocol and statistical analysis plan are available in Danish from the corresponding author upon request.
Supporting Information: Study Protocol, SAP
Time Frame: The study protocol and SAP will be available after publication and up to 5 years after the publication date.
Access Criteria: Upon reasonable request.

REFERENCES:
- [Background] Weiss J; American Academy of Pediatrics Committee on Injury, Violence, and Poison Prevention. Prevention of drowning. Pediatrics. 2010 Jul;126(1):e253-62. doi: 10.1542/peds.2010-1265. Epub 2010 May 24. PMID 20498167
- [Background] Schmidt AC, Sempsrott JR, Szpilman D, Queiroga AC, Davison MS, Zeigler RJ, McAlister SJ. The use of non-uniform drowning terminology: a follow-up study. Scand J Trauma Resusc Emerg Med. 2017 Jul 17;25(1):72. doi: 10.1186/s13049-017-0405-x. PMID 28716063
- [Background] Papa L, Hoelle R, Idris A. Systematic review of definitions for drowning incidents. Resuscitation. 2005 Jun;65(3):255-64. doi: 10.1016/j.resuscitation.2004.11.030. PMID 15919561
- [Background] Lu TH, Lunetta P, Walker S. Quality of cause-of-death reporting using ICD-10 drowning codes: a descriptive study of 69 countries. BMC Med Res Methodol. 2010 Apr 8;10:30. doi: 10.1186/1471-2288-10-30. PMID 20374660
- [Background] Steensberg J. Epidemiology of accidental drowning in Denmark 1989-1993. Accid Anal Prev. 1998 Nov;30(6):755-62. doi: 10.1016/s0001-4575(98)00028-1. PMID 9805518
- [Background] Mackie IJ. Patterns of drowning in Australia, 1992-1997. Med J Aust. 1999 Dec 6-20;171(11-12):587-90. doi: 10.5694/j.1326-5377.1999.tb123808.x. PMID 10721338
- [Background] Truhlar A, Deakin CD, Soar J, Khalifa GE, Alfonzo A, Bierens JJ, Brattebo G, Brugger H, Dunning J, Hunyadi-Anticevic S, Koster RW, Lockey DJ, Lott C, Paal P, Perkins GD, Sandroni C, Thies KC, Zideman DA, Nolan JP; Cardiac arrest in special circumstances section Collaborators. European Resuscitation Council Guidelines for Resuscitation 2015: Section 4. Cardiac arrest in special circumstances. Resuscitation. 2015 Oct;95:148-201. doi: 10.1016/j.resuscitation.2015.07.017. Epub 2015 Oct 15. No abstract available. PMID 26477412
- [Background] Venema AM, Groothoff JW, Bierens JJ. The role of bystanders during rescue and resuscitation of drowning victims. Resuscitation. 2010 Apr;81(4):434-9. doi: 10.1016/j.resuscitation.2010.01.005. Epub 2010 Feb 10. PMID 20149515
- [Background] Idris AH, Berg RA, Bierens J, Bossaert L, Branche CM, Gabrielli A, Graves SA, Handley AJ, Hoelle R, Morley PT, Papa L, Pepe PE, Quan L, Szpilman D, Wigginton JG, Modell JH; American Heart Association. Recommended guidelines for uniform reporting of data from drowning: the "Utstein style". Circulation. 2003 Nov 18;108(20):2565-74. doi: 10.1161/01.CIR.0000099581.70012.68. No abstract available. PMID 14623794
- [Derived] Breindahl N, Wolthers SA, Jensen TW, Holgersen MG, Blomberg SNF, Steinmetz J, Christensen HC; Danish Cardiac Arrest Group. Danish Drowning Formula for identification of out-of-hospital cardiac arrest from drowning. Am J Emerg Med. 2023 Nov;73:55-62. doi: 10.1016/j.ajem.2023.08.024. Epub 2023 Aug 15. PMID 37619443